CLINICAL TRIAL: NCT03180814
Title: Acute Effects of Whole Body Vibration on Autonomic Function in Healthy Young and Elderly
Brief Title: Effects of Whole Body Vibration on Autonomic Function in Healthy Young and Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Helga Cecília Muniz de Souza, Msc, Universidade Federal de Pernambuco
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WBV on autonomic function
Record Dates: First submitted 2017-03-21; First posted 2017-06-08 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Healthy; Aging

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Young Group (Active Comparator): Healthy young of both sexes between the ages of 18 and 30 years will perform a whole body vibration session
  Interventions: Other: Whole Body Vibration
- Elderly Group (Experimental): Healthy elderly of both sexes between the ages of 60 and 80 years will perform a whole body vibration session
  Interventions: Other: Whole Body Vibration

INTERVENTIONS:
Other: Whole Body Vibration — A whole body vibration session will be performed through a vibrating platform with three axes and vibration frequency set at 35 Hz. The amplitude used will be 04 mm.

SUMMARY:
Aging causes anatomical and physiological changes in the cardiovascular system and autonomic function with decline in its maximum function. This study aimed to evaluate the acute effects of whole body vibration on cardiovascular system, autonomic function and heart variability in healthy young and elderly. The investigators' hypothesis is that whole body vibration has different effects in young and elderly.

ELIGIBILITY:
Inclusion Criteria:

* Elderly individuals aged between 60 and 80 years
* Young individuals aged between 18 and 30 years
* Able to walk without assistance
* Good understanding to perform the proposed procedures
* Sedentary or low active

Exclusion Criteria:

* Body Mass Index (BMI) > 35Kg/m2
* Systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg (at rest)
* Difficulty adapting to the whole body vibration
* Smoking
* Neuromuscular or degenerative disorders
* Neurological diseases
* Cardiopulmonary comorbidities
* Cardiac arrhythmias
* Osteoarticular disorders
* Use of hormone replacement therapy
* Use medications or supplements known to affect cardiovascular parameters
* Labyrinthitis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Autonomic Function | Change from Baseline Heart rate variability at 5, 10, 15, 20 and 35 minutes
  Heart rate variability will be assessed from 3-channel holter

SECONDARY OUTCOMES:
Sympathetic modulation | Change from Baseline Sympathetic modulation at 5, 10, 15, 20 and 35 minutes
  Sympathetic modulation will be assessed from 3-channel holter
Parasympathetic modulation | Change from Baseline Parasympathetic modulation at 5, 10, 15, 20 and 35 minutes
  Parasympathetic modulation will be assessed from 3-channel holter
Sympathovagal Balance | Change from Baseline Sympathovagal balance at 5, 10, 15, 20 and 35 minutes
  Sympathovagal Balance will be assessed from 3-channel holter
Heart Rate | Change from Baseline Heart Rate at 5, 10, 15, 20 and 35 minutes
  Non-invasive measures will be assessed from 3-channel holter
Blood pressure | Change from Baseline Blood pressure at 5, 10, 15, 20 and 35 minutes
  Non-invasive measures of brachial blood pressure
Peripheral oxygen saturation | Change from Baseline Peripheral oxygen saturation at 5, 10, 15, 20 and 35 minutes
  Non-invasive measures will be assessed from pulse oximeter
Adverse effects | Change from Baseline at 20 minutes
  Adverse effects reported by volunteers

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Pernambuco, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: No